CLINICAL TRIAL: NCT06644053
Title: Exploring Locomotion Behavior of Chronic Non-Specific Low Back Pain (cNSLBP) Patients While Walking Through Apertures in Different Configurations: Influence of Environmental and Social Factors.
Acronym: PERL3
Status: Completed | Type: Observational
Sponsor: University of Rennes 2 (Other)
Responsible Party: Principal Investigator, Agathe Bilhaut, PhD, University of Rennes 2
Other Study IDs: 2023-A00870-45
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Chronic Low Back Pain (non-specific, Uncomplicated); Walking
Keywords: Chronic Low back Pain; Crossing task paradigm; ecological paradigm; Assessment; Walking; Affordance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Chronic Non-Specific Low Back Pain participants: Participants must have pain located between the thoracolumbar hinge and the lower gluteal fold, with or without pain in either leg, present for more than 12 weeks, on a daily or almost daily basis (at least 4 days out of 7).
  Interventions: Behavioral: Quantified analysis of walking during a crossing task through different horizontal openings
- Control group: Participant with no current or past chronic pain
  Interventions: Behavioral: Quantified analysis of walking during a crossing task through different horizontal openings

INTERVENTIONS:
Behavioral: Quantified analysis of walking during a crossing task through different horizontal openings — Functional test that reproduce a task of daily living

SUMMARY:
The biomechanical parameters studied in chronic non-specific low back pain (cNSLBP) patients in a locomotion task have so far focused on straight line walking. Although locomotion is primarily an automated action composed of repetitive patterns allowing movement from one place to another, walkers must respond to the environmental demands.These modifications show a flexible and adaptive approach to the constraints of the environment. This study focuses on a crossing task through different horizontal openings, varying the environmental context (two opening widths: one narrow and one wide) and the social context by placing an experimenter in the center of the two openings for some trials. The primary objective was to determine whether the cNSLBP affects the participant's decision to cross one of the two apertures as a function of the width of the aperture and the presence or absence of an experimenter. The secondary aim was twofold, firstly to study the kinematic variables of walking and secondly to assess the influence of pain perception variables on the choice of aperture crossed.

ELIGIBILITY:
Inclusion Criteria Non Specific Chronic Low Back Pain patients:

* Participants must have pain located between the thoracolumbar hinge and the lower gluteal fold, with or without pain in either leg.
* This pain must have been present for more than 12 weeks, on a daily or almost daily basis (at least 4 days out of 7)
* Participants must not be on any treatment or have been on stable analgesic treatment for at least 2 weeks prior to inclusion
* Participants must speak, read and understand French
* Participants must be between 18 and 65 years of age
* Participants must be able to understand simple commands and experimental instructions
* Participants must have normal or corrected vision
* Participants must have given informed consent to participate in the study
* Participants must be enrolled in or receiving social security benefits

Exclusion Criteria Non Specific Chronic Low Back Pain patients:

* Participants must not be pregnant or nursing mothers.
* Participants must not have cognitive or psychological impairments that are incompatible with compliance and/or understanding of the protocol
* Participants must not be unable to understand informed consent, or be under guardianship or conservatorship Subjects must not already be participating in another research protocol involving the human subject or in parallel
* Participants must not be persons deprived of liberty by judicial or administrative decision
* Participants must not be under psychiatric care
* The participants must not present neurological signs evoking a neurodegenerative disease responsible for walking disorders (parkinsonian syndrome, ...)
* The participants must not present warning signs (red flags) pointing to an underlying pathology requiring specific and/or urgent care such as
* Ongoing litigation following a work-related accident
* Pain related to a cancer diagnosis
* Associated spinal cord symptoms (pyramidal signs, coordination disorders, motor or sensory deficits, sphincter disorders, etc.)
* Pain following an infection (night sweats, fever, chills, intravenous drug abuse, immunodeficiency, recent surgery, urinary or skin infection, etc.)
* Recent or pathological fractures (traffic accidents, history of osteoporosis, chronic use of corticosteroids, advanced age, unexplained weight loss, fatigue, history of cancer, etc. )
* Vascular problems (cold feet, decreased peripheral arterial pulse, etc.)

Inclusion and Exclusion Criteria of control group :

Participants strictly meet the same inclusion and non-inclusion criteria as NSCLBP patients, but must not have ongoing chronic pain or a history of significant chronic pain (≥ 4/10 for at least 6 months). They are matched for age and gender. They must not have any pathologies that affect walking or posture. These individuals must be able to perform the studied movements without the appearance of discomfort or exaggerated fatigue.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic non-specific low back pain are recruited as part of their medical follow-up in a medical centre in France.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Critical threshold for motion adaptation | Clinical assessment at base line
  The critical threshold corresponds to the goal position at which individuals change their mode of action, i.e. the goal at which participants will cross the narrow aperture.

SECONDARY OUTCOMES:
Walking speed | Clinical assessment at base line
  Speed will calculate using the first derivative of the participant's position (location of the center of each participant at each point in time).
Clearance distance | Clinical assessment at base line
  The clearance distance corresponds to the distance between the participant and the central obstacle forming the two apertures, i.e. a pole for the condition with modified environment and a human being for the conditions with modified social factors.
Shoulder rotation | Clinical assessment at base line
  The shoulder rotation of each participant will be calculate from the horizontal coordinates of the two glenohumeral (GH) for the unobstructed straight lines and the experimental trials. The angle will be define in the horizontal plane between the GH line and the instantaneous walking direction at time where participants cross the aperture.
Phase shift between the scapular and pelvic angles | Clinical assessment at base line
  The difference between the angles of rotation of the shoulders and pelvis in the horizontal plane of each participant will be calculated from the horizontal coordinates of the displacement of the markers positioned on the two glenohumeral and on the anterior superior iliac spine for the straight-line trials with no obstacles in the path and for the experimental trials.

OTHER OUTCOMES:
Pain intensity | Clinical assessment at base line
  Pain intensity reflects the overall magnitude of the patient's perceived pain experience. The investigators will assess this variable using a visual analogue scale (VAS) in paper format. The VAS is represented by a 100 mm long horizontal line with descriptors at both ends: on the left "no pain" and on the right "worst pain imaginable". The patient must then draw a mark on the line corresponding to his or her pain experience. "0" corresponds to "no pain" and "10" corresponds to "worst pain imaginable".
Levels of anxiety and depression | Clinical assessment at base line
  Anxiety refers to fear, extreme worrying and hyperarousal symptoms. Depression refers to negative mood, loss of self-confidence, loss of motivation and pleasure. The investigators will use these measures using the Hospital Anxiety Depression Scale (HADS). This tool consists of 14 items scored from 0 to 3. Seven questions relate to anxiety (Total A) and 7 questions to the depressive dimension (Total D), resulting in two scores with a maximum total of 21 each. The higher the score, the more anxiety or depression the person has.
Pain Catastrophizing | Clinical assessment at base line
  Catastrophizing refers to the cognitive process in which anxious patients dwell on the most negative consequences and refers here to the interpretation of pain as extremely threatening. The investigators will use the Pain Catastrophizing Scale (PCS) to assess three dimensions: rumination, amplification and helplessness. This scale consists of 13 items scored from 0 (not at all) to 4 (all the time) with a maximum score of 52. The higher the score, the greater the level of catastrophisation.
Kinesiophobia | Clinical assessment at base line
  Fear of movement is characterized by pain-related fears and anxieties that often result in avoidance of movement that could cause or worsen an injury. The investigators will use the Tampa Scale Kinesiophobia (TSK). This scale consists of 17 items rated from 1 (strongly disagree) to 4 (strongly agree) with a maximum score of 68. The higher the score, the greater the level of kinesiophobia.
Psychological Inflexibility in Pain | Clinical assessment at base line
  Psychological flexibility measures psychological functioning in phase (in fusion) with the pain or whether the patient has certain degrees of freedom from it. The investigators will use the Psychological Inflexibility in Pain Scale (PIPS) allowing to assess two factors: avoidance and cognitive fusion. This scale consists of 16 items with a scale of 1 (never true) to 7 (always true). The higher the score, the greater the level of psychological inflexibility.
Fear Avoidance Beliefs | Clinical assessment at base line
  Fear and avoidance beliefs reflect patients' pain avoidance behaviors. The investigators will use the Fear Avoidance Beliefs Questionnaire (FABQ) to assess two subscales: beliefs about work and beliefs about physical activity. The questionnaire consists of 16 items scored from 0 (absolutely disagree with the sentence) to 6 (completely agree with the sentence). The maximum score for beliefs about work is 42 and the maximum score for beliefs about physical activity is 24. The higher the score, the greater the level of beliefs.
Physical functioning | Clinical assessment at base line
  Physical functioning refers to the impact on the patient's ability to perform daily physical activities necessary to meet basic needs, ranging from self-care to more complex activities that require a combination of skills. The investigators will use the Roland Morris Disability Questionnaire (RMDQ). This questionnaire has 24 items with a maximum score of 24. The higher the score, the more functional disabilities the person has.
Quality of life assessment | Clinical assessment at base line
  Quality of life refers to the impact on the physical, psychological, and social domains of health, considered as distinct domains that are influenced by a person's experiences, beliefs, expectations, and perceptions. The investigators will use the EuroQol 5 Dimension questionnaire (EQ-5D) allowing for the assessment of five dimensions: mobility, ability to care for oneself, usual work, home, and leisure activities, pain/discomfort, anxiety, and depression. Five degrees of severity in ascending order are used to assess each dimension: "no problems" to "total disability" for items that assess ability, and "no problem" to "extreme" for the other items. The higher the score, the lower the level of quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rennes 2, Rennes, France

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.